CLINICAL TRIAL: NCT00095524
Title: A Multicenter, Randomized, Double-Blind Study on the Effects of Aripiprazole in Overweight Patients Treated With Olanzapine for Schizophrenia or Schizoaffective Disorder
Brief Title: Effects of Aripiprazole in Overweight Patients Treated With Olanzapine for Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-122
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2008-05

CONDITIONS: Body Weight Change; Schizophrenia; Schizoaffective Disorder; Psychotic Disorder
Keywords: Patient weight change; changes in metabolic status
MeSH Terms: conditions — Body Weight Changes; Schizophrenia; Psychotic Disorders | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
The primary purpose of this study is to compare the affects of aripiprazole and olanzapine on weight change.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with schizophrenia or schizoaffective disorder who are currently taking olanzapine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Comparison of weight change from baseline to Week 16 in patients with schizophrenia or schizoaffective disorder treated with aripiprazole or olanzapine

SECONDARY OUTCOMES:
Assessment of metabolic laboratory measures

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (32):
- United States (23):
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Anaheim, California
  - Local Institution, Cerritos, California
  - Local Institution, Garden Grove, California
  - Local Institution, National City, California
  - Local Institution, San Diego, California
  - Local Institution, New Britain, Connecticut
  - Local Institution, North Miami, Florida
  - Local Institution, Augusta, Georgia
  - Local Institution, Macon, Georgia
  - Local Institution, Hoffman Estates, Illinois
  - Local Institution, Louisville, Kentucky
  - Local Institution, Glen Burnie, Maryland
  - Local Institution, Haverhill, Massachusetts
  - Local Institution, Worcester, Massachusetts
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Brooklyn, New York
  - Local Institution, Nashville, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, DeSoto, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Wauwatosa, Wisconsin
- Brazil (7):
  - Local Institution, Goibnia, Goiás
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Botucatu, São Paulo
  - Local Institution, Sao Paulo - Sp, São Paulo
  - Local Institution, São Paulo, São Paulo
- United Kingdom (2):
  - Local Institution, Exeter, Devon
  - Local Institution, Birmingham, West Midlands

REFERENCES:
- [Derived] Newcomer JW, Campos JA, Marcus RN, Breder C, Berman RM, Kerselaers W, L'italien GJ, Nys M, Carson WH, McQuade RD. A multicenter, randomized, double-blind study of the effects of aripiprazole in overweight subjects with schizophrenia or schizoaffective disorder switched from olanzapine. J Clin Psychiatry. 2008 Jul;69(7):1046-56. doi: 10.4088/jcp.v69n0702. PMID 18605811